CLINICAL TRIAL: NCT01603719
Title: Safety and Efficacy of an Infant Starter Formula With Prebiotics (GOS) and a Higher Content of Beta-palmitate on Stool Characteristics, Food Tolerance, Calcium Uptake, and Incidence of Infectious Disease in the First Year of Life
Brief Title: Efficacy and Safety of an Infant Formula With Milkfat and Prebiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Waldkrankenhaus Protestant Hospital, Spandau (Other)
Responsible Party: Principal Investigator, Antonia Nomayo, MD, MD, Waldkrankenhaus Protestant Hospital, Spandau
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EWK-001
Record Dates: First submitted 2012-05-15; First posted 2012-05-23 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Infections; Stool Flora; Stool Biochemistry; Constipation; Food Intolerance
Keywords: infant formula; prebiotics; beta-palmitate; stool flora; bifidogenic
MeSH Terms: conditions — Infections; Constipation; Food Intolerance | interventions — Prebiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Formula (No Intervention): Standard formula with no supplementation
- experimental formula (Experimental): infant formula with higher beta-palmitate and supplemented GOS
  Interventions: Dietary Supplement: new infant formula with prebiotics and beta-palmitate

INTERVENTIONS:
Dietary Supplement: new infant formula with prebiotics and beta-palmitate — experimental infant formula as sole source of nutrition over first 12 weeks of life
  Arms: experimental formula

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of a new infant starter formula with added prebiotics (GOS) and with a fat blend rich in beta-palmitate.

DETAILED DESCRIPTION:
An experimental infant formula with added prebiotics (GOS) and with a higher content of palmitic acid esterified in beta-position is to be tested in a double-blinded randomized controlled trial.

The addition of prebiotics to an infant formula should favor growth of a beneficial bifidogenic intestinal flora and have positive effects on immunity, promote softer stool formation and short chain fatty acid content in the stools. Higher proportion of beta-palmitic acid esterified in 2nd position of the triglyceride should reduce formation of fatty acid-calcium soaps in the stools and promote calcium and fat absorption in the gut, therfor reduce symptoms of constipation and colics.

ELIGIBILITY:
Inclusion Criteria:

* healthy term neonates
* gestational age 37 to 42 weeks
* birth weight 10th to 90th percentile (Voigt reference)
* infants being exclusively formula-fed at enrollment

Exclusion Criteria:

* infants with high risk of atopic disease due to family history
* congenital disorder or syndrome with need for special diet / impairment of growth
* antibiotic medication prior to enrollment

Max Age: 10 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
number of gastrointestinal infections | within first year of life

SECONDARY OUTCOMES:
proportion of bifidobacteria on total stool bacteria | after 6 and 12 weeks intervention
number of infectious episodes (gastrointestinal, respiratory, fever episodes) | within first year of life
anthropometric parameters (gain in weight, length, head circumference) | after 6 weeks, after 12 weeks intervention
symptoms of food intolerance, constipation, colics | after 6 weeks, 12 weeks intervention
  number of episodes with colics, vomiting, abdominal bloating, intestinal gas; stool frequency, stool consistency, constipation
stool biochemistry (calcium-fatty acid soaps, short chain fatty acids content in the stools) | after 6 weeks, 12 weeks intervention
atopic manifestation | within 1st year of life
  incidence atopic dermatitis
erythrocytes´ fatty acid profile | after 6 weeks intervention
  palmitic acid, linolic acid, alpha-linoleic acid, AA, DHA, EPA etc content (erythrocytes membrane)
calcium absorption | after 6 weeks, 12 weeks intervention
  urinary calcium-creatinin ratio, serum alkaline phosphatase

CONTACTS AND LOCATIONS:
Overall Officials: Frank Jochum, MD, Principal Investigator — Waldkrankenhaus Protestant Hospital, Spandau
Locations (1):
- Evangelisches Waldkrankenhaus Spandau, Berlin, Germany

REFERENCES:
- [Derived] Lambidou M, Alteheld B, Fimmers R, Jochum F, Nomayo A, Stehle P. Impact of an Infant Formula Containing a Novel Fat Blend (Cow's Milk Fat, Fish and Vegetable Oil) and Prebiotics on Stool Fatty Acid Soaps and Erythrocyte Fatty Acid Profiles in Full-Term Healthy Newborns. Ann Nutr Metab. 2021;77(3):138-145. doi: 10.1159/000515705. Epub 2021 Apr 30. PMID 33934094
- [Derived] Nomayo A, Schwiertz A, Rossi R, Timme K, Foster J, Zelenka R, Tvrdik J, Jochum F. Infant formula with cow's milk fat and prebiotics affects intestinal flora, but not the incidence of infections during infancy in a double-blind randomized controlled trial. Mol Cell Pediatr. 2020 Jul 2;7(1):6. doi: 10.1186/s40348-020-00098-1. PMID 32613402